CLINICAL TRIAL: NCT01080430
Title: Short-term and Long-term Effects of the Rotational Maneuver in Patients With Chronic Vestibular Imbalance
Brief Title: Effects of a Vestibular Rehabilitation Maneuver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Day General Hospital. (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Nayer Rassaian, Professor / Doctor, Shahid Beheshti University of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: DGH-VR02
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Vertigo
Keywords: vestibular; vertigo; rehabilitation; rotation; balance
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: rehabilitation maneuver — rotation in the direction of the weak vestibular response, every 3-7 days over a period of a month. Each rotation lasts about 2 minutes and a total of 3-7 rotations are used per session.
  Other Names: rotatory maneuver

SUMMARY:
Rotational maneuver is a vestibular rehabilitation method, performed in a supervised manner. Using a rotating chair, subjects are rotated towards the opposite direction of dominant side in order to inhibit this side and simultaneously, stimulate the subordinate side. We propose that the rehabilitative effect is the result of a decrease in the vestibular imbalance, mainly due to a decrease in the response of the dominant vestibular side. Previously, we have shown the short-term effects of this maneuver on patients with recent onset vestibular imbalance. In the present study, we investigated the long-term effects of the rotational maneuver in patients with a history of peripheral vestibular vertigo for at least one year, originally confirmed by clinical tests. Our results show a significant improvement which lasted for >4 weeks after the end of rehabilitation (i.e., the last time tested). Moreover, there seems to be a relationship between the decrease in DP values and a decrease in subjective symptoms. We propose that this maneuver can be used as an effective method for both short- and long-term rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* History of vertigo for at least one year
* Not under drug therapy for vertigo
* directional preponderance >10% measured by electronystagmography during rotation test

Exclusion Criteria:

* severe vertigo
* intolerance to rotation
* previously diagnosed for a central pathology (e.g., neuroma)
* previously diagnosed with a fluctuating vestibular disorder (e.g., Menier's)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Directional preponderance (DP) | Every 3-7 days for one month
  It provides an objective measure of vestibular asymmetry (percentage) in response to rotation. Eye movements are measured by electronystagmography during head rotations to the right and to the left. DP (%) is calculated by the equation: 100 x (max eye velocity for rightward rotations - max eye velocity for left rotations) / (max eye velocity for rightward rotations + max eye velocity for left rotations). Values below 10% are considered normal.

SECONDARY OUTCOMES:
Subjective sense of a decrease in imbalance and dizziness. | every 3-7 days for one month
  Patients report the intensity and frequency of their symptoms as a measure of subjective improvement on a scale of 1 - 10, with 10 representing the most improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Nayer Rassaian, MD, PhD, Principal Investigator — Shaheed Beheshti University
Locations (1):
- Vestibular and auditory center of Day General Hospital, Tehran, Iran

REFERENCES:
- [Derived] Sadeghi NG, Sabetazad B, Rassaian N, Sadeghi SG. Rebalancing the Vestibular System by Unidirectional Rotations in Patients With Chronic Vestibular Dysfunction. Front Neurol. 2019 Jan 22;9:1196. doi: 10.3389/fneur.2018.01196. eCollection 2018. PMID 30723455